CLINICAL TRIAL: NCT05805319
Title: Randomized Dietary Intervention to Improve Fiber Intake in Patients With Non-small Cell Lung Cancer Treated With Immune Checkpoint Inhibitor Therapy
Brief Title: Dietary Intervention for NSCLC Patients Treated With ICI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22.261
Record Dates: First submitted 2023-02-15; First posted 2023-04-10 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Diet; Fiber Intake; Immune checkpoint inhibitor therapy; NSCLC; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-center randomized trial in patients with non-small cell lung cancer (NSCLC) treated with immune checkpoint inhibition. Patients will receive standard-of-care immune checkpoint inhibitor (ICI) therapy alone or in combination with a dietary intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients in the control arm will complete the dietary survey without dietary intervention or counselling from a dietician. Control group will have dietary survey and 24-hour recall survey at baseline, at 6 weeks, and at 12 weeks relative to ICI initiation.
- Intervention Group (Experimental): Patients in the intervention arm will complete a dietary survey and be counselled on increasing their total fiber intake. Intervention group will have dietary survey and 24-hour recall survey at baseline, at 6 weeks, and at 12 weeks relative to ICI initiation.
  Interventions: Other: increasing total fiber intake

INTERVENTIONS:
Other: increasing total fiber intake — Patients in the intervention arm will complete a dietary survey and be counselled on increasing their total fiber intake.
  Arms: Intervention Group

SUMMARY:
This is a single-center randomized trial in patients with non-small cell lung cancer (NSCLC) treated with immune checkpoint inhibition. Patients will receive standard-of-care immune checkpoint inhibitor (ICI) therapy alone or in combination with a dietary intervention.

DETAILED DESCRIPTION:
Nutritionist-guided dietary intervention in patients with NSCLC treated with ICI can improve patients' fiber intake.

Intervention:

After 1:1 randomization, patients in the intervention arm will complete a dietary survey and be counselled on increasing their total fiber intake. Patients in the control arm will complete the dietary survey without dietary intervention or counselling from a dietician. Both the intervention and control groups will have dietary survey and 24-hour recall survey at baseline, at 6 weeks, and at 12 weeks relative to ICI initiation.

Details of Dietary Intervention: Nutritionists will perform a standard evaluation, which includes a nutritional assessment of the patient's current dietary intake. The intervention will follow Canada Food Guide's recommendations (https://food-guide.canada.ca) for healthy eating with the addition of personalized recommendations on how to increase foods rich in dietary fiber. Recommendations may include food substitutions to food equivalent options that are richer in fiber, such as exchanging low fiber white bread to whole wheat bread for an increase in 3g of fiber per slice. Recommendations may also include adding fiber-rich foods and Mediterranean meals or snacks, with a supporting document highlighting inexpensive options such as frozen vegetables and fruit, rolled oats, canned or dried pulses, whole wheat pasta or whole grain rice. Patients will receive a document that lists food sources of fiber as well as generalized recommendations on how to incorporate them into daily eating habits. They will be counselled how to read food labels to identify fiber content of packaged foods. On average, participants will be encouraged to choose or add foods richer in fiber to achieve 5-10 g of fiber per meal with snacks containing 3-5 g of fiber. They will not be asked to track the grams of fiber they eat, the nutritionist will measure their fiber intake and will adjust her recommendations in order to achieve 25 g of fiber or more. Although there is no tolerable upper limit set for fiber, the nutritional intervention will aim to avoid an excess fiber intake (60-70g) to prevent displacement of other nutrients and a negative impact on nutritional adequacy of the diet. The current recommended adequate intake of fiber set for adults is based on approximately >25 g per day. Participants will be encouraged to increase their fiber in a gradual step-wise manner (approximately 5-10 g maximum per day) to limit possible digestive side effects from too rapid of an introduction. For patients with diarrhea, a known possible side effect of immunotherapy, they will be advised to select food sources that are rich in soluble fiber rather than insoluble fibers.

ELIGIBILITY:
Inclusion Criteria:

* Signed, informed consent
* Age 18 years or older
* Confirmed histological diagnosis of non-small cell lung cancer (NSCLC); Treatment with standard-of-care ICI
* Ability to eat solid foods

Exclusion Criteria:

* Severe dietary allergies (e.g. shellfish, nuts, seafood)
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in the intervention arm (nutritionist intervention) with total daily fiber intake of >=25g/day compared to the control arm (no nutritionist intervention). | 12 weeks
  Proportion of patients in the intervention arm (nutritionist intervention) with total daily fiber intake of >=25g/day compared to the control arm (no nutritionist intervention).

SECONDARY OUTCOMES:
Proportion of patients in the intervention arm (nutritionist intervention) with improved Panagiotakos MedDietScore (defined by a score higher than 26.25 on 55 or an increase of 10 points)) compared to the control arm (no nutritionist intervention). | 12 weeks
  By assessing the change in global dietary habits as measured by the Panagiotakos MedDietScore.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Routy, MD,PhD, Principal Investigator — CHUM
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No